CLINICAL TRIAL: NCT03874039
Title: Exploratory Study of Sweat Cytokines and Insensible Gas Losses From Skin in Healthy Normal Adults and Patients With Atopic Dermatitis
Brief Title: Sweat and Gas Sensor for Healthy Skin and Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Shuai (Steve) Xu, Principal Investigator, Northwestern University
Other Study IDs: SX09092018
Record Dates: First submitted 2019-01-29; First posted 2019-03-14 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Healthy Adults; Atopic Dermatitis; Wearables; Sweat Sensor; Gas Sensor
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Adults: Healthy adults with no prior diagnosis of atopic dermatitis
  Interventions: Device: Gas sensor; Device: Sweat Sensor
- Atopic Dermatitis: Adults with prior diagnosis of Atopic Dermatitis from board certified dermatologist
  Interventions: Device: Gas sensor; Device: Sweat Sensor

INTERVENTIONS:
Device: Gas sensor — The gas sensor is an airtight gas capsule attached with a floating solid phase microextraction (SPME) tube. SPME uses a fiber coated with a nontoxic liquid (polymer), and a nontoxic solid (sorbent). The fiber coating extracts the compounds from the gas being released from the skin. Only the glass sample is in contact with the skin.
Device: Sweat Sensor — The sweat sensor is a soft, flexible device that rests on the skin and collects secreted sweat through capillary action. The device is held in place by medical-grade acrylic adhesive film.

SUMMARY:
Pilot study of a wearable gas and sweat skin sensor

DETAILED DESCRIPTION:
The objective of this study is exploratory and deploys two wearable sweat and gas sensors which detect the composition of sweat proteins and volatile gases emitted from the skin in healthy subjects and patients with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Subjects willing and able to comply with requirements of the protocol
* Healthy adults or subjects with atopic dermatitis

Exclusion Criteria:

* Age <18 years old
* Subjects unwilling and able to comply with requirements of the protocol
* History of skin allergy to medical adhesive tape
* History of heat stroke, heat related or exercise related
* Non-English speaking subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults and adults with prior diagnosis of atopic dermatitis from made by board certified dermatologist
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Evaluation of gas exudates | 20 minutes
  Evaluation of protein contents from gas exudates from the skin
Evaluation of sweat proteins | 20 minutes
  Evaluation of protein contents from sweat from the skin

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xu, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States